CLINICAL TRIAL: NCT04536818
Title: Outcomes After Laparotomy for Penetrating Abdominal Trauma: A Cohort Study From a Tertiary Trauma Hospital in South Africa
Brief Title: Outcomes After Laparotomy for Penetrating Abdominal Trauma
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Andreas Älgå, Principal Investigator, Karolinska Institutet
Other Study IDs: TraumaLapCohort
Record Dates: First submitted 2020-08-21; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Penetrating Abdominal Trauma
MeSH Terms: interventions — Laparotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Time to surgery ≤12 hours: Waiting time to surgery ≤12 hours from hospital presentation.
  Interventions: Procedure: Laparotomy
- Time to surgery >12 hours: Waiting time to surgery >12 hours from hospital presentation.
  Interventions: Procedure: Laparotomy

INTERVENTIONS:
Procedure: Laparotomy — Exploratory laparotomy.

SUMMARY:
The purpose of this study is to evaluate outcomes of adult patients hospitalised due to penetrating abdominal trauma at a tertiary trauma hospital in South Africa. Our primary objective is to study the association between waiting time to surgery and outcome (mortality, complications, and length of hospital stay) in normotensive patients treated with laparotomy for penetrating abdominal trauma.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are admitted due to penetrating abdominal injuries, irrespective of injury mechanism, time from injury and prior treatment.
* Patients that are treated with laparotomy.

Exclusion Criteria:

* Patients that are admitted due to blunt trauma or combinations of blunt and penetrating trauma.
* Patients who are dead on arrival.
* Patients that are only re-admitted during the study period, i.e. patients that received primary treatment by TBH before study initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Tygerberg Academic Hospital, Cape Town, South Africa.
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Death | Through study completion, an average of 2 weeks
  In-hospital death.

SECONDARY OUTCOMES:
Complications | Through study completion, an average of 2 weeks
  Complications according to the Clavien-Dindo classification.
Length of stay | Through study completion, an average of 2 weeks
  Length of hospital stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Tygerberg Academic Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No